CLINICAL TRIAL: NCT01422655
Title: Accuracy of Transcutaneous Bilirubin Determinations in Neonates: The Effect of Gestational Age, Time and Site of Measurement
Brief Title: Transcutaneous Bilirubinometry in Neonates
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Fouzas Sotirios, Pediatrician, Neonatal Intensive Care Unit, University Hospital of Patras, University of Patras
Other Study IDs: TcB_Patr_2011
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Neonatal Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: To assess the accuracy of transcutaneous bilirubin (TcB) measurements in neonates, in relation to gestational age (GA), time (postnatal hour) and site (forehead, sternum, knee) of measurements.

Hypothesis: Using (or combining) different sites for TcB determination might improve the accuracy of TcB in relation to the time of measurement and the GA of the neonate.

Methods: The study will include neonates >32 weeks' gestation cared for in the well-baby nursery and NICU of the University Hospital of Patras, from September to December 2011. Data such as sex, gestational age, gestation and perinatal information, mother's and infant's ABO group and Rh, G6PD deficiency, Coombs test, type of delivery and complications, birthweight, postnatal medications and interventions, type and volume of feeding, and extension of jaundice, will be collected.

TcB measurements will be performed using the BiliCheck bilirubinometer (according to the standard protocol) at 3 different sites: forehead, sternum and knee. Total serum bilirubin (TSB) values will be obtained using the heel stick technique, and measurements will be performed by a direct spectrophotometric device (Unistat bilirubinometer, Richert, Depew, NY). The accuracy of the device has been validated previously. TSB measurements will be performed within 5 minutes of the TcB measurements.

At each occasion TcB measurements (3), the corresponding TSB value, the time of measurement (postnatal hours), and the actual weight will be noted.

Statistics: The agreement between TcB and TSB values will be assessed using the Bland-Altman % method. The independent and joint effects of GA and time of measurement on bias will be evaluated by multivariate regression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Born at the University Hospital of Patras
2. GA >32 weeks
3. Parental consent to participate

Exclusion Criteria:

1. Under phototherapy
2. Congenital infections
3. Chromosomal abnormalities
4. Congenital abnormalities
5. Hepatic dysfunction

Max Age: 120 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term and preterm neonates from birth to 120 postnatal hours
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Accuracy characteristics of TcB as compared to TSB | Tcb vs TSB measurements at any time from birth to 120 postnatal hours
  TcB measurements performed at 3 different sites (forehead, sternum, knee)will be compared with the corresponding TSB value. The agreement between TcB and TSB values will be assessed using the Bland-Altman % method. The effect of gestational age and time of measurement (postnatal hour)on TcB bias will be explored by multivariate regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Fouzas, MD, Principal Investigator — Neonatal Intensive Care Unit, University Hospital of Patras; Anastasia Varvarigou, Prof, Study Director — Neonatal Intensive Care Unit, University Hospital of Patras; Eugenia Panagiotopoulou, MD, Principal Investigator — Neonatal Intensive Care Unit, University Hospital of Patras
Locations (1):
- Neonatal Intensive Care Unit, University Hospital of Patras, Pátrai, Greece